CLINICAL TRIAL: NCT06685094
Title: Cross-cultural Adaptation, Translation and Validation of the Assessment Scales of the Upper and Lower Limbs, Pain, Autonomy and Quality of Life for Use in the Albanian-speaking Population
Brief Title: Translation and Validation of the Upper and Lower Limbs, Pain, Autonomy and Quality of Life Scales in Albanian
Status: Recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Orges Lena, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: CE052107
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Pain; Autonomy; Healthy; Upper Limb Injury; Lower Limb Injury
MeSH Terms: conditions — Musculoskeletal Pain; Arm Injuries; Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cross-cultural adaptation will be performed according to the internationally recommended methodology, using the following guidelines: translation, back-translation; revision by a committee, questionnaire diffusion and data collection and analyzing.

The psychometric properties will be evaluated by administering the questionnaire to approximately 300 participants. Reliability will be estimated through stability and homogeneity assessment

DETAILED DESCRIPTION:
The assessment scales of the upper and lower limbs, pain, autonomy and quality of life for use in the Albanian-speaking population are as follow:

1. Adaptation, validation and test-retest reliability of upper limbs scales as: Disabilities of the arm, shoulder and hand questionnaire (DASH), MAYO Elbow score, oxford Elbow score, patent-rated tennis elbow evaluation, shoulder pain and disability index (SPADI), Simple Shoulder Test (SST) and Upper Limp Functional Index (ULFI).
2. Adaptation, validation and test-retest reliability of lower limb scales as: Oxford Hip Score, Motricity Index and Trunk Control Test in Albanian language.
3. Adaptation, validation and test-retest reliability of health scales and autonomy: Functional Ambulation Category (FAC), Fear-Avoidance Beliefs Questionnaire (FABQ), Graded Chronic Pain Scale (GCPS),Motor Assessment Scale (MAS), Stroke rehabilitation Assessment of movement (STREAM), Hospital Anxiety and Depression Scale (HADS), Headache Impact Test (HIT6), Leeds Assessment of Neuropathic Symptoms and Signs pain scale (LANSS), Instrumental activities of daily living scale (IADL), health status questionnaire (EQ-5D-5L), Social Responsiveness Scale (SRS), short portable mental status questionnaire (SPMSQ), Tampa Skale Kinesiophobia, Ankle--Hindfoot Scale (AOFAS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* articular and muscular pain
* back pain
* presence of rheumatologic symptoms
* functional misbalance
* scoliosis
* musculoskeletal disorders

Exclusion Criteria:

* no native albanian language
* severe trauma to the lumbar spine or hip(s)
* tumor
* metabolic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Albanian patients whom seeking care for articular and muscular pain.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Adaptation, validation and test-retest reliability of upper limbs scales | 7 days
  validation of the scales for the: disabilities of the arm, shoulder and hand questionnaire (DASH), MAYO Elbow score, oxford Elbow score, patent-rated tennis elbow evaluation, shoulder pain and disability index (SPADI), Simple Shoulder Test (SST) and Upper Limp Functional Index (ULFI).
Adaptation, validation and test-retest reliability of lower limb scales | 7 days
  validation of the scales for the: Oxford Hip Score, Motricity Index and Trunk Control Test in Albanian language.
Adaptation, validation and test-retest reliability of health scales and autonomy | 7 days
  validation of : Functional Ambulation Category (FAC), Fear-Avoidance Beliefs Questionnaire (FABQ), Graded Chronic Pain Scale (GCPS),Motor Assessment Scale (MAS), Stroke rehabilitation Assessment of movement (STREAM), Hospital Anxiety and Depression Scale (HADS), Headache Impact Test (HIT6), Leeds Assessment of Neuropathic Symptoms and Signs pain scale (LANSS), Instrumental activities of daily living scale (IADL), health status questionnaire (EQ-5D-5L), Social Responsiveness Scale (SRS), short portable mental status questionnaire (SPMSQ), Tampa Skale Kinesiophobia, Ankle--Hindfoot Scale (AOFAS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

CONTACTS AND LOCATIONS:
Locations (1):
- Jasemin Todri, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No